CLINICAL TRIAL: NCT05287802
Title: The Efficacy of Balance and Proprioception Exercises in Patients With Knee Osteoarthritis: a Randomized Controlled Study
Brief Title: The Efficacy of Balance and Proprioception Exercises in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BI1422
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis; Balance; Distorted; Proprioceptive Disorders
MeSH Terms: conditions — Osteoarthritis, Knee; Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: This study was planned to compare the effects of isometric strengthening exercises plus balance and proprioception exercises performed by two different methods with isometric strengthening exercises alone. This was a single-center randomized trial with 3 parallel arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patients, the outcome assessor, care provider physicians, and the statistician were blinded to allocation. The supervising physician was not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biodex Training (BT) group (Active Comparator): Biodex Balance System features a platform that can move simultaneously in the anteroposterior (AP) or medio-lateral (ML) direction in 12 different levels of stability within a 20-degree range of inclination, as well as a locked position for static environments. For this platform, 1 represents the least stable level and 12 represents the most stable level. Interactive, game-like training modes are provided with the on-screen grid and score-keeping functions. Patients in the BT group performed exercises with the Balance SystemTM SD once a day, three days a week for 10 weeks under the physicians' supervision. Furthermore this group received closed kinetic chain exercises (CKCE) in addition to their own exercise program, which was applied in exactly the same way. The CKCE were performed in three sets of 10 repetitions with five seconds rest between each exercise. The exercises consisted of mini-squats, wall sits, and lunges.
  Interventions: Other: Balance and proprioception exercises
- Classical balance training group (CT group) (Active Comparator): Patients in the CT group completed the exercise program once a day and three days a week during the 10-week period under the physicians' supervision. The exercises consisted of standing on one leg, tandem walking (heel-to-toe), balance board exercises, Romberg exercise, backward walking, and side-to-side stepping exercises. The total duration of these exercises was 20-30 minutes. Furthermore this group also received CKCE in addition to their own exercise program, which was applied in exactly the same way. The CKCE were performed in three sets of 10 repetitions with five seconds rest between each exercise. The exercises consisted of mini-squats, wall sits, and lunges.
  Interventions: Other: Balance and proprioception exercises
- Control group (Active Comparator): Isometric home exercises, which can be considered the most basic and feasible strengthening program, were selected to compare the effects they had when added to the intervention groups and administered alone. All patients in the study performed isometric exercises for the quadriceps and hamstrings at home once a day, three days a week for 10 weeks. The exercises were performed as 10 repetitive cycles of six-second contractions and two-second rest periods. All patients were given a daily exercise chart to mark the home program, and adherence to the exercises was monitored weekly by telephone call.
  Interventions: Other: Home exercises program

INTERVENTIONS:
Other: Balance and proprioception exercises — Balance and proprioception exercises using two different methods (classical balance training and Biodex) in addition to strengthening exercises
  Arms: Biodex Training (BT) group; Classical balance training group (CT group)
Other: Home exercises program — Isometric exercises for the quadriceps and hamstrings at home
  Arms: Control group

SUMMARY:
This study aime to investigate the effects of balance and proprioception exercises using two different methods (classical balance training and Balance System™ SD) in addition to strengthening exercises on dynamic balance, pain, functional status and quality of life in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
It is known that knee OA leads to a decrease in proprioception and balance disturbances. Falls due to balance disorders often occur during dynamic activities such as walking and stair climbing. Therefore, correction of balance disorders is of great importance to prevent falls and associated fractures in the elderly population, in which knee OA is common. In addition, loss of proprioception in the knee joint, muscle weakness, and balance disorders are also known to contribute to the development of knee OA itself. Therefore, treatment of balance disorders may also slow the progression of the disease. This study was planned to compare the effects of isometric strengthening exercises plus balance and proprioception exercises performed by two different methods with isometric strengthening exercises alone. This is a single-center randomized trial with 3 parallel arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they had a knee OA diagnosis according to the American College of Rheumatology (ACR) diagnostic criteria, had suffered from knee pain for at least six months, had radiologically verified bilateral knee OA of grade II or III according to the Kellgren-Lawrence classification and had not previously participated in a regular exercise program.

Exclusion Criteria:

* Patients who had undergone knee surgery, who had received hyaluronic acid or corticosteroid injections into the knee within six months, and patients with conditions that might affect balance were excluded from the study.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | Baseline
  The postural stability test, was performed with the following parameters: Duration: 20 seconds, Stability level: 8, and Stance: two legs. The value of overall stability index (OSI) is obtained by calculating the standard deviations of the degrees of inclination with respect to the zero point (locked position). Higher values indicate poorer equilibrium.
Dynamic balance | 10th week
  The postural stability test, was performed with the following parameters: Duration: 20 seconds, Stability level: 8, and Stance: two legs. The value of overall stability index (OSI) is obtained by calculating the standard deviations of the degrees of inclination with respect to the zero point (locked position). Higher values indicate poorer equilibrium.
Dynamic balance | Baseline
  The modified Clinical Test of Sensory Interaction and Balance (mCTSIB).The entire test is performed with the platform in the locked position. The test consists of 4 conditions: Condition 1: eyes open firm surface, Condition 2: eyes closed firm surface, Condition 3: eyes open dynamic (foam) surface, and Condition 4: eyes closed dynamic (foam) surface. The firm and dynamic surface tests assess static and dynamic balance, respectively. The conditions under which visual data are blocked are designed to detect even minor balance disturbances caused by the sensorimotor system. The sway index obtained as a result of the test represents the average position of the patient's center of mass relative to the center of the platform. Higher values indicate poorer balance. mCTSIB Condition-3, and mCTSIB Condition-4 dynamic balance assessment tests were used to assess dynamic balance.
Dynamic balance | 10th week
  The modified Clinical Test of Sensory Interaction and Balance (mCTSIB).The entire test is performed with the platform in the locked position. The test consists of 4 conditions: Condition 1: eyes open firm surface, Condition 2: eyes closed firm surface, Condition 3: eyes open dynamic (foam) surface, and Condition 4: eyes closed dynamic (foam) surface. The firm and dynamic surface tests assess static and dynamic balance, respectively. The conditions under which visual data are blocked are designed to detect even minor balance disturbances caused by the sensorimotor system. The sway index obtained as a result of the test represents the average position of the patient's center of mass relative to the center of the platform. Higher values indicate poorer balance. mCTSIB Condition-3, and mCTSIB Condition-4 dynamic balance assessment tests were used to assess dynamic balance.

SECONDARY OUTCOMES:
Pain score | Baseline
  Patients' pain scores at night, at rest, and during movement were measured using visual analogue scale (VAS) (0-10 cm; 0 indicates no pain and 10 indicates severe pain).
Pain score | 10th week
  Patients' pain scores at night, at rest, and during movement were measured using visual analogue scale (VAS) (0-10 cm; 0 indicates no pain and 10 indicates severe pain).
Physical function | Baseline
  Physical function was assessed using the 30-second chair stand test (30CST) , which is recommended by the Osteoarthritis Research Society International (OARSI). Patients sit in a chair with the knees bent slightly more than 90 degrees and the feet on the floor at an angle behind the knees. While arms are crossed in front of the chest, patients stand up with lower limbs fully extended and sit back down with full contact to the chair. The movement of standing up and sitting down is counted as one cycle. The number of cycles during the 30-second period is recorded. Increasing values indicate good performance.
Physical function | 10th week
  Physical function was assessed using the 30-second chair stand test (30CST) , which is recommended by the Osteoarthritis Research Society International (OARSI). Patients sit in a chair with the knees bent slightly more than 90 degrees and the feet on the floor at an angle behind the knees. While arms are crossed in front of the chest, patients stand up with lower limbs fully extended and sit back down with full contact to the chair. The movement of standing up and sitting down is counted as one cycle. The number of cycles during the 30-second period is recorded. Increasing values indicate good performance
Physical function | Baseline
  Physical function was assessed using the 40-meter fast-paced walk test (40-m-FPWT) , which is recommended by the Osteoarthritis Research Society International (OARSI). Two cones are used to mark the start and stop lines of a 10-meter walkway. Patients are asked to walk as fast as they can along the walkway without running, and then turn around four times, and the total time recorded. Decreasing values indicate good performance
Physical function | 10th week
  Physical function was assessed using the 40-meter fast-paced walk test (40-m-FPWT) , which is recommended by the Osteoarthritis Research Society International (OARSI). Two cones are used to mark the start and stop lines of a 10-meter walkway. Patients are asked to walk as fast as they can along the walkway without running, and then turn around four times, and the total time recorded. Decreasing values indicate good performance
Quality of life (QoL) | Baseline
  QoL of patients was assessed using the QoL subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS). The KOOS consists of five subscales assessing pain, other symptoms, activities of daily living, sports and leisure time, and QoL. Each question is scored on a five-point scale ranging from 0 to 4. Scores close to 100 represent good outcomes, while scores close to 0 represent poor outcomes
Quality of life (QoL) | 10th week
  QoL of patients was assessed using the QoL subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS). The KOOS consists of five subscales assessing pain, other symptoms, activities of daily living, sports and leisure time, and QoL. Each question is scored on a five-point scale ranging from 0 to 4. Scores close to 100 represent good outcomes, while scores close to 0 represent poor outcomes

CONTACTS AND LOCATIONS:
Overall Officials: BUGRA INCE, MD, Principal Investigator — Bozyaka Training and Research Hospital; ALTINAY GOKSEL KARATEPE, MD, Study Director — University of Health Sciences Izmır Faculty, Bozyaka Training and Research Hospital
Locations (1):
- Izmir Bozyaka Research and Training Hostpital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
upon request

REFERENCES:
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Anwer S, Alghadir A, Brismee JM. Effect of Home Exercise Program in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. J Geriatr Phys Ther. 2016 Jan-Mar;39(1):38-48. doi: 10.1519/JPT.0000000000000045. PMID 25695471
- [Background] Niino N, Tsuzuku S, Ando F, Shimokata H. Frequencies and circumstances of falls in the National Institute for Longevity Sciences, Longitudinal Study of Aging (NILS-LSA). J Epidemiol. 2000 Apr;10(1 Suppl):S90-4. doi: 10.2188/jea.10.1sup_90. PMID 10835834
- [Background] Khan SJ, Khan SS, Usman J, Mokhtar AH, Abu Osman NA. Effects of different foot progression angles and platform settings on postural stability and fall risk in healthy and medial knee osteoarthritic adults. Proc Inst Mech Eng H. 2018 Feb;232(2):163-171. doi: 10.1177/0954411917750409. Epub 2017 Dec 28. PMID 29283019
- [Background] Jan MH, Lin CH, Lin YF, Lin JJ, Lin DH. Effects of weight-bearing versus nonweight-bearing exercise on function, walking speed, and position sense in participants with knee osteoarthritis: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Jun;90(6):897-904. doi: 10.1016/j.apmr.2008.11.018. PMID 19480863